CLINICAL TRIAL: NCT00427843
Title: The Influence of a Home Program of Hip Abductor Exercises on Gait Parameters and Muscle Strength in Persons With Knee Osteoarthritis
Brief Title: The Influence of Hip Strengthening Exercises on Walking Patterns and Muscle Strength in Persons With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Elsie Culham, PhD, School of Rehabilitation Therapy, Queen's University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REH-324-06
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; gait; muscle strength; hip; exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise Home-Based Program (Experimental): Patients with knee OA will be taught a home-based exercise program for the hip abductor muscles during the initial visit. The exercise program will be performed 3 times per week for 8 weeks.
  Interventions: Behavioral: home exercise program for the hip abductor muscles

INTERVENTIONS:
Behavioral: home exercise program for the hip abductor muscles — All patients with knee OA will be taught a home-based exercise program for the hip abductor muscles during the initial visit. Patients will be instructed in the following program: contraction of the gluteus medius muscle during functional activities (gait, stepping sideways up on a step and standing on one leg); and side lying isotonic hip abduction exercises using graded resistance elastic bands positioned around the distal thighs.
  The program will be performed 3 times per week for 8 weeks and subjects will record exercise frequency and level of resistance on exercise calendars. Follow-up visits will occur at the end of week 1 and week 4 for review and progression of exercises. A telephone follow-up call will occur for support and participants will be encouraged to call with any questions or concerns.

SUMMARY:
The purpose of this study is to determine the influence of a home program of exercises for the hip muscles which support the pelvis on walking patterns and hip muscle strength in people with knee osteoarthritis. Following a hip muscle strengthening program, we hypothesize that participants with knee osteoarthritis will demonstrate decreased loading at the knee joint during walking and greater strength of the hip muscles.

DETAILED DESCRIPTION:
Knee osteoarthritis is a common age-related impairment that may progress to cause significant pain and physical disability. Excessive loading at the knee joint is believed to contribute to the progression of knee osteoarthritis. The hip joint and surrounding muscles have been shown to influence the amount of stress occurring at the knee joint during walking. In particular, the hip abductor muscles may have an effect on the knee joint by controlling the position of the pelvis and/or by acting as lateral stabilizers for the knee.

Research suggests that the function of the hip muscles during walking may be decreased in people with knee osteoarthritis and that greater loads may be placed on the knee joint as a result. Thus, interventions aimed at strengthening the hip abductor muscles may be effective for reducing stress on the arthritic knee and slowing the rate of progression of knee osteoarthritis.

The design of the study is a two-group pretest-posttest design using an untreated control group. Thirty-five individuals with medial compartment knee osteoarthritis will be recruited through newspaper advertisements and from the practices of orthopedic surgeons in Kingston, Ontario. Each participant with knee osteoarthritis will be matched with an asymptomatic volunteer for age (+/- 5 years), height (+/- 5 cm), mass (+/- 5 kg) and gender. Participants in the control group will have no clinical or radiographic diagnosis of knee or hip osteoarthritis or rheumatoid arthritis and no history of hip or knee trauma or pain.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 40 years
* self-reported pain in the knee(s) for most days of the month
* at least some difficulty in daily function due to knee osteoarthritis
* radiographic evidence of knee osteoarthritis or documented evidence of cartilage loss in the knee by arthroscopy surgery or magnetic resonance imaging.

Exclusion Criteria:

* corticosteroid injection into either knee within the previous three months
* other significant medical problems (including significant heart disease, stroke and active treatment for cancer) that would prevent participants from being able to perform a hip exercise program or to participate in tests of walking performance and hip muscle strength
* known osteoarthritis or previous trauma affecting one or both hips
* previous replacement of any joint in the lower extremities.
* receiving rehabilitation services for knee osteoarthritis or performing a hip strengthening program at the time of testing
* participants who have had a dual-energy x-ray absorptiometry (DEXA) for bone density analysis or more than one x-ray of the chest, abdomen or hip in the past 6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Walking variables: hip and knee abductor and adductor moments | baseline and after 8 weeks
Muscle strength measures: isometric and isokinetic peak torque measures for the hip abductor and adductor muscles | baseline and after 8 weeks

SECONDARY OUTCOMES:
Radiographs: lower limb frontal plane alignment measures - limb alignment in degrees; grading of knee osteoarthritis severity (total score out of 13) | baseline
Speed of performance on the Five-Times-Sit-to-Stand Test | baseline and after 8 weeks
Total score on the WOMAC pain subscale and the WOMAC physical function subscale | baseline and after 8 weeks
Total score obtained for the physical activity scale (PASE) | baseline and after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elsie G. Culham, PhD, Study Director — Queen's University
Locations (1):
- School of Rehabilitation Therapy, Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Sled EA, Khoja L, Deluzio KJ, Olney SJ, Culham EG. Effect of a home program of hip abductor exercises on knee joint loading, strength, function, and pain in people with knee osteoarthritis: a clinical trial. Phys Ther. 2010 Jun;90(6):895-904. doi: 10.2522/ptj.20090294. Epub 2010 Apr 8. PMID 20378679